CLINICAL TRIAL: NCT01201304
Title: Comparison of Methods for the Delivery of Interoceptive Exposure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Wyoming (Other)
Responsible Party: Principal Investigator, Brett Deacon, Associate Professor of Psychology, University of Wyoming
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEstudyUW
Record Dates: First submitted 2010-09-09; First posted 2010-09-14 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Anxiety Sensitivity
Keywords: Anxiety sensitivity; Panic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interoceptive exposure (Experimental): Repeated trials of voluntary hyperventilation intended to reduce fears of arousal-related body sensations.
  Interventions: Behavioral: Standard exposure; Behavioral: Enhanced exposure; Behavioral: Intensive exposure
- Expressive writing (Placebo Comparator): Expectancy control intervention.
  Interventions: Behavioral: Expressive writing

INTERVENTIONS:
Behavioral: Standard exposure — Three 60-second trials of hyperventilation, each followed by diaphragmatic breathing, cognitive reappraisal, and prolonged rest until body sensations have subsided.
  Arms: Interoceptive exposure
Behavioral: Enhanced exposure — Three 60-second trials of hyperventilation, each followed by a 15-second rest period and cognitive reappraisal.
  Arms: Interoceptive exposure
Behavioral: Intensive exposure — Minimum of eight 60-second hyperventilation trials, each followed by 15-second rest period and cognitive reappraisal. Trials continue until participants rate the probability that their most feared outcome will occur as less than 5% on a 0% to 100% scale.
  Arms: Interoceptive exposure
Behavioral: Expressive writing — Individuals randomized to the expressive writing control group will receive a rationale for why writing about emotional issues helps resolve the fear of body sensations. These participants will then be asked to spend the next 25 minutes writing about past emotional issues. Participant writings are confidential and will not be viewed by the experimenter.
  Arms: Expressive writing

SUMMARY:
This study compares the relative efficacy of three methods of delivering interoceptive exposure for the reduction of elevated anxiety sensitivity. The interventions vary according to their intensity and use of coping strategies during exposure. An expressive writing intervention serves as an expectancy control.

DETAILED DESCRIPTION:
Cognitive-behavioral theories posit that panic attacks and panic disorder are the product of inaccurate beliefs about the dangerousness of arousal-related body sensations such as heart palpitations, dizziness, and shortness of breath. Individuals with panic disorder often misinterpret these anxiety symptoms as likely to lead to health catastrophes such as a heart attack, stroke, suffocation, or insanity. Effective psychological treatment aims to correct such misinterpretations by helping individuals learn that their anxiety-related body sensations are not dangerous.

One treatment procedure used to accomplish this goal is "interoceptive exposure," or the deliberate evocation of anxiety-related body sensations via exercises such as hyperventilation, spinning in a swivel chair, or running in place. By demonstrating that the experience of anxiety-related body sensations does not lead to physical catastrophes, interoceptive exposure exercises help individuals learn not to fear their own anxiety symptoms. Indeed, this procedure is considered an essential ingredient in evidence-based psychological treatment of panic disorder.

Despite the established therapeutic value of interoceptive exposure, little is known about how to optimally deliver this procedure. In the most clinically tested panic disorder treatment package, individuals engage in three, minute-long trials of interoceptive exposure exercises such as hyperventilation, with each trial followed by the use of diaphragmatic breathing and a rest period until all anxiety-related body sensations have subsided. However, there are theoretical reasons to question the effectiveness of this method. For example, encouraging individuals to use controlled breathing to "manage" their sensations appears incompatible with the notion that anxiety-related body sensations are harmless. Similarly, the instruction to wait until one's body sensations have subsided to begin the next interoceptive exposure trial suggests that intense body sensations are to be avoided. For these reasons, many practitioners conduct interoceptive exposure in a more intensive manner in which individuals experience feared body sensations in a prolonged fashion, without attempting to suppress or avoid them, until they learn that the sensations are harmless. Despite the theoretical appeal of this latter approach, no studies have examined the effects of delivering interoceptive exposure in this manner. Indeed, very little is known about the effects of different methods of delivering interoceptive exposure on fear of arousal-related body sensations. Accordingly, the present study aims to test the effectiveness of different methods of delivering interoceptive exposure with the goal of generating recommendations for the optimal treatment of panic disorder and other clinical problems associated with the fear of anxiety-related body sensations.

ELIGIBILITY:
Inclusion Criteria:

* Score > 21 on Anxiety Sensitivity Index - Revised Fear of Respiratory Symptoms Subscale.

Exclusion Criteria:

* Seizures
* Hypertension
* Heart problems
* Pregnancy
* Asthma
* Other health conditions exacerbated by intense exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Fear of Anxiety-Related Body Sensations | Immediately following the single-session intervention
  Anxiety Sensitivity Index - Revised Concerns Subscale (12 items)
Fear of Anxiety-Related Body Sensations | One week after single-session intervention
  Anxiety Sensitivity Revised - Respiratory Concerns Subscale (12 items)

SECONDARY OUTCOMES:
Hypervigilance to anxiety-related body sensations | One week after the single-session intervention
  Body Vigilance Scale (4 items)
Beck Anxiety Inventory | One week after the single-session intervention
  Beck Anxiety Inventory (21 items)
Peak Anxiety During a Symptom Induction Task | Immediately following the single-session intervention
  Peak anxiety ratings during prolonged straw breathing
Peak Anxiety During a Symptom Induction Task | One week after the single-session intervention
  Peak anxiety ratings during prolonged straw breathing

CONTACTS AND LOCATIONS:
Overall Officials: Brett Deacon, Ph.D., Principal Investigator — University of Wyoming
Locations (1):
- University of Wyoming, Laramie, Wyoming, United States